CLINICAL TRIAL: NCT05826821
Title: Circulating Biomarkers of Fibrosis and Cardiovascular Disease in Patients With Heart Failure With Preserved Ejection Fraction - Analysis of Samples Collected as Part of the PIROUETTE Trial
Brief Title: Biomarkers in HF: Circulating Biomarkers of Fibrosis and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B01793; 320856 (Registry Identifier: IRAS ID)
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Heart Failure with Preserved Ejection Fraction; Myocardial Fibrosis; Myocardial Extracellular Volume; Pirfenidone
MeSH Terms: conditions — Heart Failure | interventions — pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pirfenidone: Pirfenidone 801mg capsule by mouth, three times a day (target dose) for 12 months
  Interventions: Drug: Pirfenidone
- Placebo: Placebo capsule by mouth, three times a day (target dose) for 12 months

INTERVENTIONS:
Drug: Pirfenidone — Intervention drug
  Groups: Pirfenidone

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) represents one of the largest unmet needs in cardiovascular medicine. Heart muscle scarring (myocardial fibrosis) is a key HFpEF disease mechanism and represents an important therapeutic target.

Myocardial fibrosis can be measured non-invasively using the cardiovascular magnetic resonance imaging (MRI) extracellular volume (ECV) technique. However, some patients cannot undergo MRI scanning, and it is expensive. Circulating biomarkers in the blood that are sensitive to changes in myocardial fibrosis would represent an attractive cheaper and accessible alternative.

This study aims to assess baseline levels of, and longitudinal change in, circulating biomarkers relating to fibrosis and cardiovascular disease in gifted samples from PIROUETTE trial participants, and evaluate the relationship between the biomarkers, anti-fibrotic treatment response and other study measurements.

DETAILED DESCRIPTION:
Myocardial fibrosis, is a key HFpEF disease mechanism and represents an important therapeutic target.

Myocardial fibrosis is caused by excess secretion of collagen and other large molecules within the heart. Several of these molecules can be detected and measure in blood serum, thereby acting as non-invasive markers of myocardial fibrosis. Examples include, but are not limited to, precursors of type I and type 3 collagen.

In addition, gut microorganisms produce imidazole propionate (ImP), which can be detected in blood samples. This molecule has previously been associated with cardiovascular disease and heart failure and the investigators hypothesise that it may also be associated with myocardial fibrosis.

These circulating biomarkers of fibrosis are a cheaper and more accessible alternative for measurement of cardiac fibrosis compared to cardiovascular MRI ECV technique.

This study will investigate the association between circulating biomarkers of fibrosis, gut microbiome function and cardiovascular disease in samples from PIROUETTE.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male or female; aged 40 years or older.
* HF, defined as one symptom present at the time of screening, and one sign present at the time of screening or in the previous 12 months. Symptoms and signs are defined as:
* Symptoms: dyspnoea on exertion, orthopnoea or paroxysmal nocturnal dyspnoea Signs: peripheral oedema, crackles on chest auscultation post-cough, raised jugular venous pressure or chest x-ray demonstrating pleural effusion, pulmonary congestion, or cardiomegaly
* Left Ventricular Ejection Fraction (LVEF) > 45% at Visit 0, (any local LVEF measurement made using echocardiography or CMR).
* BNP ≥ 100 pg/ml or NTproBNP ≥ 300 pg/ml recorded at Visit 0. For patients in atrial fibrillation on Visit 0 ECG, BNP > 300pg/ml or NTproBNP > 900 pg/ml at Visit 0.
* Myocardial fibrosis, defined as Extracellular Matrix (ECM) volume > 27% by CMR at Visit 0.

Exclusion Criteria:

* Myocardial infarction, coronary artery bypass graft surgery or percutaneous coronary intervention within the previous 6 months.
* Probable alternative cause of patient's HF symptoms that in the opinion of the investigator primarily accounts for patient's dyspnoea such as significant pulmonary disease, anaemia or obesity. Specifically, patients with the below are excluded:

Severe chronic obstructive pulmonary disease (COPD) (i.e., requiring home oxygen, chronic nebuliser therapy, or chronic oral steroid therapy), or Haemoglobin < 9 g/dl, or Body mass index (BMI) > 55 kg/m2. Known pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy.

Clinically significant congenital heart disease. Presence of severe valvular heart disease. Atrial fibrillation or flutter with a resting ventricular rate > 100 bpm. Any medical condition, which in the opinion of the Investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.

* Severe renal dysfunction at Visit 0, defined as estimated Glomerular Filtration Rate (eGFR) <30 mL/min (using Chronic Kidney Disease Epidemiology Collaboration Equation (CKD-EPI) calculation), or end-stage renal disease requiring dialysis.
* History of severe hepatic impairment or liver dysfunction at Visit 0, defined as total bilirubin above the upper limit of normal (ULN) (excluding patients with Gilbert's syndrome), aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 times the ULN or alkaline phosphatase >2.5 times the ULN.
* Prolonged corrected QT interval, defined as a corrected QT interval >500 msec on ECG using Bazett formula.
* Known hypersensitivity to any of the components of the investigational medicinal product (IMP).
* Use of other investigational drugs at the time of enrolment, or within 30 days or 5 half-lives of enrolment, whichever is longer.
* Fluvoxamine use within 28 days of Visit 0.
* Contraindication to MRI scanning or gadolinium-based contrast agent
* Pregnancy, lactation or planning pregnancy. Women of childbearing capacity are required to have a negative serum pregnancy test before treatment, must agree to pregnancy tests at study visits as defined in the Section 7.2.5 and must agree to maintain highly effective contraception during the study and for 3 months thereafter. Similarly male participants with female partners of childbearing potential must agree to maintain highly effective contraception during the study and for 3 months thereafter.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with preserved ejection fraction and myocardial fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Circulating biomarkers of myocardial fibrosis | 12 months
  Examples include procollagen type I C-terminal propeptide (PICP) and collagen type I C-terminal telopeptide (CITP) in micrograms per litre

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided